CLINICAL TRIAL: NCT02586701
Title: Effects of a Supervised Versus Non-supervised Exercise Program on Adherence and Functional Outcomes in Colorectal Cancer Patients
Brief Title: Supervised Versus Non-supervised Exercise on Adherence and Functional Outcomes in Colorectal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franco Carli (Other)
Responsible Party: Sponsor-Investigator, Franco Carli, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MM123
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation Plus (Active Comparator): Patients in this group will be enrolled in a multimodal program before surgery involving supervised exercise, nutrition counseling and relaxation strategies. Supervised exercise is provided once a week for four weeks before surgery as well as during the hospital stay post surgery. Patients are to continue with a home-based exercise program for 8 weeks after discharge.
  Interventions: Other: Prehabilitation Plus
- Rehabilitation (No Intervention): Patients in this group are provided with in-hospital supervised exercises with a kinesiologist post surgery until discharge. Patients, upon discharge are provided with a home-based exercise program, nutritional counseling and relaxation strategies for 8 weeks.

INTERVENTIONS:
Other: Prehabilitation Plus — Supervised exercise program and home-based exercise program.
  Arms: Prehabilitation Plus

SUMMARY:
Investigation into prehabilitation by increasing the supervision of exercise in patients undergoing colorectal resection for cancer and comparing with patients involved in a rehabilitation group receiving exercise after surgery.

DETAILED DESCRIPTION:
The aims of this research project are the following:

To determine to what extent a structured multimodal prehabilitation regimen, which includes aerobic and resistance exercise, nutritional supplementation and psychological coping strategies, initiated before surgery, and continued while in hospital and after surgery, optimizes the recovery of functional walking capacity following colorectal resection for cancer.

To understand which measures of immediate surgical recovery are sensitive to prehabilitation interventions and predict change in later outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* referred electively for resection of malignant, non metastasized, colorectal lesions.
* French or English speaking

Exclusion Criteria:

* ASA class 4-5
* co-morbid medical, physical and mental conditions (e.g. dementia, disabling orthopedic and neuromuscular disease, psychosis)
* cardiac abnormalities
* severe end-organ disease such as cardiac failure (New York Heart Association classes I-IV), COPD, renal failure (creatinine > 1.5mg/dl, and hepatic failure ALT and AST > 50% over the normal range)
* Sepsis
* Morbid obesity (BMI > 40)
* Anemia (hematocrit < 30%, haemoglobin < 10g/dl, albumin < 25mg/dl).

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Test (6MWT) | up to 8 weeks after surgery
  Change in functional walking capacity will be assessed throughout the study according to the 6-Minute Walk Test (6MWT). The 6MWT evaluates the ability of an individual to maintain a moderate level of physical activity over a time period reflective of the activities of daily living. Subjects are instructed to walk back and forth, in a 20 m stretch of hallway, for six-minutes, at a pace that would make them tired by the end of the walk; encouragement and feedback are given according to published guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Carli, MD, Study Chair — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Gillis C, Li C, Lee L, Awasthi R, Augustin B, Gamsa A, Liberman AS, Stein B, Charlebois P, Feldman LS, Carli F. Prehabilitation versus rehabilitation: a randomized control trial in patients undergoing colorectal resection for cancer. Anesthesiology. 2014 Nov;121(5):937-47. doi: 10.1097/ALN.0000000000000393. PMID 25076007
- [Background] Mayo NE, Feldman L, Scott S, Zavorsky G, Kim DJ, Charlebois P, Stein B, Carli F. Impact of preoperative change in physical function on postoperative recovery: argument supporting prehabilitation for colorectal surgery. Surgery. 2011 Sep;150(3):505-14. doi: 10.1016/j.surg.2011.07.045. PMID 21878237
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub3. PMID 37162250
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2022 May 19;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub2. PMID 35588252
- [Derived] Gillis C, Fenton TR, Sajobi TT, Minnella EM, Awasthi R, Loiselle SE, Liberman AS, Stein B, Charlebois P, Carli F. Trimodal prehabilitation for colorectal surgery attenuates post-surgical losses in lean body mass: A pooled analysis of randomized controlled trials. Clin Nutr. 2019 Jun;38(3):1053-1060. doi: 10.1016/j.clnu.2018.06.982. Epub 2018 Jul 9. PMID 30025745